CLINICAL TRIAL: NCT05586347
Title: Relationship Between Perioperative Carotid Blood Flow Monitoring and Cerebral Function Protection in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hongwei Shi, Head of the anesthesia department, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: hongweishi
Record Dates: First submitted 2022-10-13; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Bypass Grafting; Cardiopulmonary Bypass
MeSH Terms: interventions — Nicardipine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group N (Experimental): Nicardipine was infused after initiation of CPB
  Interventions: Drug: Nicardipine
- group C (Placebo Comparator): Give the same volume of normal saline
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: Nicardipine — Nicardipine 0.2-0.5μg/(kg·min) was infused at the beginning of CPB.
  Other Names: Astellas Pharmaceuticals (China) Co., LTD；Sinopharm approved number J20160048/ Registration number H20160015
  Arms: group N
Other: normal saline — It has the same capacity as group N。
  Other Names: Hunan Kelun Pharmaceutical Co., LTD；Sinopharm approved H43020456
  Arms: group C

SUMMARY:
Postoperative cognitive dysfunction (POCD) is a common complication of cardiac surgery, mainly manifested as mental confusion, anxiety, personality change and memory impairment, which seriously affects the quality of life of patients after surgery.Attention should be paid to the protection of neurological function in patients undergoing cardiac surgery during perioperative period.Nicardipine can selectively act on coronary arteries and cerebral vessels, increase coronary artery and cerebral blood flow, relieve coronary heart disease angina pectoris, protect brain tissue.The cerebral protective effect of nicardipine on cardiovascular surgery under CPB deserves further clinical study.About 15-20% of cardiac output (CO) in healthy adults is allocated to the brain , and cerebral blood flow is supplied by bilateral internal carotid artery (ICA) and vertebral artery (VA), among which ICA provides about 70%-80% of cerebral perfusion flow .However, the location of the internal carotid artery is superficial, the anatomical variation is less, and the ultrasonic Doppler technique is portable and simple to measure. It may be of certain clinical value to use the ultrasonic detection technology to quickly evaluate the cerebral perfusion during the perioperative period, and to early detect and avoid the intraoperative brain function injury.

DETAILED DESCRIPTION:
Patients who were scheduled to undergo open-heart surgery under cardiopulmonary bypass were randomly divided into nicardipine group (group N) and normal saline control group (group C) by the digital table method. Group N was pumped with nicardipine 0.2-0.5μg/(kg·min) after CPB, while group C was given the same volume of normal saline. The basic hemodynamic parameters, rScO2, BIS, maximum systolic velocity of internal carotid artery (PSV-ICA), end-diastolic velocity of internal carotid artery (EDV-ICA), diameter of internal carotid artery (D-ICA), internal carotid artery blood flow (Q-ICA) and cerebral blood flow ratio (CBF/CO) were observed and recorded in the two groups at each time point ), cerebrovascular resistance (CVR) and the concentration of NSE, a biomarker of brain injury.The following hypothesis is proposed: during CPB, pump nicardipine can dilate the internal carotid artery and cerebral arterioles, increase cerebral blood flow, improve cerebral oxygen supply, and reduce the risk of postoperative cognitive dysfunction（POCD）.

ELIGIBILITY:
Inclusion Criteria:

* 1: Age 60-80

  2: ASA Ⅱ-Ⅲ, NYHAⅠ-Ⅲ, EF ≥50%

  3: CABG under cardiopulmonary bypass

Exclusion Criteria:

* 1: Patients who had second heart surgery

  2: Patients with intellectual disabilities, deafness or other impairments in normal communication

  3: Previous neurosurgical procedures and history of cerebral infarction

  4: cancer

  5: Patients with moderate to severe carotid artery stenosis before operation

  6: Patients with obvious abnormal liver and kidney function affecting drug metabolism

  7: Patients taking psychotropic drugs

  8: Alcoholism, drug addiction, drug dependence

  9: The cardiopulmonary bypass time was greater than 120 minutes

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Internal carotid blood flow | Before induction of anesthesia
  Blood flow through the internal carotid artery was measured per minute by ultrasound
Internal carotid blood flow | Surgical skin excision
  Blood flow through the internal carotid artery was measured per minute by ultrasound
Internal carotid blood flow | During cardiopulmonary bypass
  Blood flow through the internal carotid artery was measured per minute by ultrasound
Internal carotid blood flow | After cardiopulmonary bypass
  Blood flow through the internal carotid artery was measured per minute by ultrasound

SECONDARY OUTCOMES:
Regional cerebral oxygen | Before induction of anesthesia
  After the forehead skin is degreased and dried with alcohol,attach the NIRS probe.
Regional cerebral oxygen | Surgical skin excision
  After the forehead skin is degreased and dried with alcohol,attach the NIRS probe.
Regional cerebral oxygen | During cardiopulmonary bypass
  After the forehead skin is degreased and dried with alcohol,attach the NIRS probe.
Regional cerebral oxygen | After cardiopulmonary bypass
  After the forehead skin is degreased and dried with alcohol,attach the NIRS probe.
Mini-mental State Examination scale score | 1 day before surgery
  Illiteracy group (no education) less than 17 points, primary school group (education ≤6 years) less than 20 points, secondary school or above group (education > 6 years) less than 24 points, the above is normal.
Mini-mental State Examination scale score | 7 days after surgery.
  Illiteracy group (no education) less than 17 points, primary school group (education ≤6 years) less than 20 points, secondary school or above group (education > 6 years) less than 24 points, the above is normal.
Neuron specific endase | Before induction of anesthesia
  3ml arterial blood was collected and centrifuged. The plasma was stored in a refrigerator at -70℃ for measurement, and the concentration of NSE was determined by ELISA.
Neuron specific endase | 2 hours after surgery.
  3ml arterial blood was collected and centrifuged. The plasma was stored in a refrigerator at -70℃ for measurement, and the concentration of NSE was determined by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: hongwei shi, Study Director — Director of anesthesiology department of Nanjing First Hospital
Locations (1):
- Hongwei Shi, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No